CLINICAL TRIAL: NCT00326911
Title: A Phase II, Randomized, Open-Label Study of Cetuximab and Bevacizumab Alone or in Combination With Fixed-Dose Rate Gemcitabine as First-Line Therapy of Patients With Metastatic Adenocarcinoma of the Pancreas
Brief Title: Cetuximab and Bevacizumab With or Without Gemcitabine to Treat Metastatic Pancreatic Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The planned enrollment was 130 patients and the study was halted prematurely due to lack of efficacy in both arms. Enrolled patients continued treatment.
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Chief Medical Officer, ImClone LLC
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CP02-0555
Record Dates: First submitted 2006-05-15; First posted 2006-05-17 (Estimated); Results first posted 2009-12-04 (Estimated); Last update posted 2011-05-25 (Estimated); Status verified 2011-05

CONDITIONS: Metastatic Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Cetuximab; Bevacizumab; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- cetuximab + bevacizumab + gemcitabine (Experimental): Cetuximab 400 mg/m2 weekly (over 120 minutes) on day 1 of cycle 1 with subsequent weekly infusions of 250 mg/m2 (over 60 minutes), followed by bevacizumab 10 mg/kg (over 60 minutes) on day 1 and repeated every 2 weeks, and gemcitabine 1000 mg/m2/minute over 100 minutes weekly x 3 of 4 weeks. All medications will be administered by intravenous infusion on the same day. The order of study drug administration will be cetuximab, bevacizumab, and gemcitabine. On day 1 of cycle 1, one hour must elapse between administration of cetuximab and bevacizumab.
  Interventions: Biological: cetuximab; Biological: bevacizumab; Drug: gemcitabine
- cetuximab + bevacizumab (Active Comparator): Cetuximab 400 mg/m2 weekly (over 120 minutes) on day 1 of cycle 1 with subsequent weekly infusions of 250 mg/m2 (over 60 minutes), followed by bevacizumab 10 mg/kg (over 60 minutes) on day 1 and repeated every 2 weeks. Both medications will be administered by intravenous infusion on the same day. The order of study drug administration will be cetuximab and bevacizumab. On day 1 of cycle 1, one hour must elapse between administration of cetuximab and bevacizumab.
  Interventions: Biological: cetuximab; Biological: bevacizumab

INTERVENTIONS:
Biological: cetuximab — I.V. infusion of 400 mg/m2 (over 120 minutes) on day 1 of cycle 1
  Other Names: Erbitux®
Biological: bevacizumab — 10 mg/kg (over 60 minutes) on day 1 and repeated every 2 weeks.
  Other Names: Avastin®
Drug: gemcitabine — 1000 mg/m2 administered intravenously at 10 mg/m2/minute over 100 minutes weekly x 3 of 4 weeks.
  Other Names: Gemzar®
  Arms: cetuximab + bevacizumab + gemcitabine
Biological: cetuximab — I.V.infusions of 250 mg/m2 (over 60 minutes) weekly
  Other Names: Erbitux®

SUMMARY:
Eligible patients with metastatic pancreatic cancer will be treated with dual agent monoclonal antibody consisting of cetuximab and bevacizumab alone or in combination with gemcitabine

ELIGIBILITY:
Inclusion Criteria:

* The patient has provided signed written informed consent.
* The patient is ≥18 years of age.
* The patient has histologically or cytologically-confirmed pancreatic adenocarcinoma not amenable to curative treatment with surgery or has documented or suspected extrapancreatic metastases.
* The patient has either (a) measurable disease as defined by Response Evaluation Criteria in Solid Tumors Version 1.0 (RECIST) or (b) non-measurable disease with an elevated baseline CA19-9 level (≥2 x the upper limit of normal [ULN]).
* The patient's Eastern Cooperative Oncology Group (ECOG) performance status is ≤2.
* The patient has adequate hematologic function as defined by an absolute neutrophil count (ANC) ≥1500/mm3 and a platelet count ≥100,000/mm3 obtained within 2 weeks prior to the first dose of study medication.
* The patient has adequate hepatic function as defined by a total bilirubin ≤2.0 mg/dL and transaminases ≤5.0 x ULN obtained within 2 weeks prior to the first dose of study medication.
* The patient has adequate renal function as defined by serum creatinine ≤2.0 x ULN and urine dipstick for proteinuria ≤1+ obtained within 2 weeks prior to the first dose of study medication. If urine dipstick is ≥2+, then a 24-hour urine for protein must demonstrate < 1000 mg of protein in 24 hours to allow participation in the study. Urinalysis is also acceptable.
* If the patient is on full-dose anticoagulation therapy (eg, warfarin or low molecular weight [LMW] heparin), the following criteria must be met:

  * The patient has an in-range International Normalized Ratio ([INR]usually between 2 and 3) on a stable dose of oral anticoagulant or be on a stable dose of LMW heparin
  * The patient has no active bleeding or pathological condition that carries a high risk of bleeding (e.g., tumor involving major vessels or known varices)
* If the patient is not on full-dose anticoagulation therapy, the following criteria must be met:

  * The patient has adequate coagulation function as defined by INR ≤1.5
  * The patient has a partial thromboplastin (PTT) ≤ULN obtained within 2 weeks prior to the first dose of study medication
* If a woman, the patient agrees to use an accepted and effective method of contraception (hormonal or barrier methods, abstinence) prior to study entry and for the duration of the study. If a male and sexually active, the patient agrees to use effective contraception.
* The patient is accessible for treatment and follow-up. Patients enrolled in this trial must be treated at the participating center.

Exclusion Criteria:

* Endocrine tumors or lymphoma of the pancreas
* Known brain metastases
* Prior therapy with an epidermal growth factor receptor (EGFR) inhibitor or vascular endothelial growth factor (VEGF) inhibitor
* Prior chemotherapy, hormonal therapy, or radiation therapy for advanced pancreatic cancer, patients who received chemotherapy and/or radiation therapy in the adjuvant setting will be eligible as long as the adjuvant therapy was completed >6 months prior
* Concurrent malignancy other than non-melanomatous skin cancer or carcinoma in situ of the cervix
* Concurrent treatment with other anti-cancer therapy, including other chemotherapy, immunotherapy, hormonal therapy, radiotherapy, chemoembolization, or targeted therapy
* Ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations
* History of arterial thrombotic events within 9 months
* History of uncontrolled hypertension (>150/100 mmHg) not on a stable regimen of anti-hypertensive therapy
* History of significant bleeding events or upper or lower gastrointestinal bleeding within 9 months
* History of gastrointestinal perforation within 12 months
* Serious non-healing wound ulcer, bone fracture, or major surgical procedure with 28 days
* If a woman, is pregnant or lactating
* An employee of the investigator or study center as well as family members of the employees

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2006-05; Primary Completion 2008-10 (Actual); Study Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: E-mail: ClinicalTrials@ ImClone.com, Study Chair — Eli Lilly and Company
Locations (15):
- United States (15):
  - ImClone Investigational Site, Jonesboro, Arkansas
  - ImClone Investigational Site, San Francisco, California
  - ImClone Investigational Site, Stamford, Connecticut
  - ImClone Investigational Site, Miami, Florida
  - ImClone Investigational Site, Orlando, Florida
  - ImClone Investigational Site, Atlanta, Georgia
  - ImClone Investigational Site, Augusta, Georgia
  - ImClone Investigational Site, Marietta, Georgia
  - ImClone Investigational Site, Metairie, Louisiana
  - ImClone Investigational Site, Billings, Montana
  - ImClone Investigational Site, Concord, North Carolina
  - ImClone Investigational Site, Philadelphia, Pennsylvania
  - ImClone Investigational Site, Charleston, South Carolina
  - ImClone Investigational Site, Arlington, Texas
  - ImClone Investigational Site, Dallas, Texas

REFERENCES:
- [Derived] Ko AH, Youssoufian H, Gurtler J, Dicke K, Kayaleh O, Lenz HJ, Keaton M, Katz T, Ballal S, Rowinsky EK. A phase II randomized study of cetuximab and bevacizumab alone or in combination with gemcitabine as first-line therapy for metastatic pancreatic adenocarcinoma. Invest New Drugs. 2012 Aug;30(4):1597-606. doi: 10.1007/s10637-011-9691-8. Epub 2011 Jun 1. PMID 21629990

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited from a population of pancreatic cancer patients treated at investigational centers.
Pre-assignment Details: Prior chemotherapy, hormonal therapy, radiation therapy in the adjuvant setting were allowed, provided that the last date of therapy was at least 6 months prior to randomization.
Groups:
- Cetuximab + Bevacizumab + Gemcitabine: Cetuximab 400 mg/m2 weekly (over 120 minutes) on day 1 of cycle 1 with subsequent weekly infusions of 250 mg/m2 (over 60 minutes), followed by bevacizumab 10 mg/kg (over 60 minutes) on day 1 and repeated every 2 weeks, and gemcitabine 1000 mg/m2/minute over 100 minutes weekly x 3 of 4 weeks. Both medications will be administered by intravenous infusion on the same day. The order of study drug administration will be cetuximab, bevacizumab, and gemcitabine. On day 1 of cycle 1, one hour must elapse between administration of cetuximab and bevacizumab.
Period: Overall Study
Arm/Group | Cetuximab + Bevacizumab + Gemcitabine | Cetuximab + Bevacizumab
Started | 30 (This number reflects all randomized patients.) | 31 (This number reflects all randomized patients.)
Completed | 29 (This number reflects all treated patients.) | 29 (This number reflects all treated patients.)
Not Completed | 1 | 2
Not completed — Hospitalization prior to treatment | 0 | 1
Not completed — Physician decision prior to treatment | 1 | 0
Not completed — Withdrawal by subject prior to treatment | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cetuximab + Bevacizumab + Gemcitabine | Cetuximab + Bevacizumab | Total
Number analyzed (Participants) | 30 | 31 | 61
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 18 | 18 | 36
  >=65 years | 12 | 13 | 25
Age Continuous [Mean (Standard Deviation); unit: years] | 62.7 (11.6) | 62.2 (11.4) | 62.4 (11.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 15 | 26
  Male | 19 | 16 | 35
Region of Enrollment [Number; unit: participants]
  United States | 30 | 31 | 61

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival (PFS)
Description: Progression-free survival is the time from randomization until the date of progressive disease (PD) or death from any cause whichever is first reported. Patients who die without a reported prior progression were considered to have progresssed on the day of their death. Patients who did not progress were censored at the day of their last tumor assessment.
Time Frame: Time from randomization to disease progression or death from any cause (Range: 0 -10 months)
Population: The PFS was based on the modified Intent-to-Treat (mITT) population, which included any patient who enrolled, was randomized, and received any quantity of study drug.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cetuximab + Bevacizumab + Gemcitabine | Cetuximab + Bevacizumab
Number analyzed (Participants) | 29 | 29
months | 3.55 [2.00 to 5.59] | 1.91 [1.81 to 2.76]

2. Secondary Outcome: Overall Survival (OS)
Description: This measure is defined as the time from randomization to the date of death due to any cause. Survival of living patients or those who lost to follow-up were censored on the last date the patients were known to be alive.
Time Frame: Survival information was collected continuously every 3 months after completion of therapy and/or follow-up (range: 1-19 months).
Population: The overall survival was based on the mITT population.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Cetuximab + Bevacizumab + Gemcitabine | Cetuximab + Bevacizumab
Number analyzed (Participants) | 29 | 29
Months | 5.41 [3.84 to 6.74] | 4.17 [2.69 to 8.74]

3. Secondary Outcome: The Number of Patients With a Best Overall Response of Either a Complete Response (CR) or Partial Response (PR)
Description: The best overall response is the number of patients with a best overall response of CR or PR, as classifed by the investigator according to the RECIST guidelines. A CR is the disappearance of all target lesions and a PR is at least a 30% decrease in the sum of the longest diameters of target lesions, taking as reference the baseline sum longest diameter.
Time Frame: Tumor evaluations were performed every 8 weeks while on cetuximab therapy until PD or recurrence. Patients with a PR or CR had a confirmatory tumor assessment no less than 4 weeks after the initial evaluation.
Population: The best overall response was based on the mITT population for those patients who either had a CR or PR.
Measure: Number; unit: Participants
Arm/Group | Cetuximab + Bevacizumab + Gemcitabine | Cetuximab + Bevacizumab
Number analyzed (Participants) | 29 | 29
Participants | 4 [3.9 to 31.7] | 0 [0.1 to 17.8]

4. Secondary Outcome: Percentage of Patients With Carbohydrate Antigen 19-9 (CA19-9) Response at End of Cycle 2 in Patients With Elevated Baseline Values (Equal or Greater Than 2 x Upper Limit of Normal).
Description: CA19-9 is a tumor marker for pancreatic cancer and the level usually increases as the disease is progressing. The CA19-9 response was the percentage of patients whose CA19-9 level was declining, stable or increasing < 10% compared with baseline, divided by the total patients with elevated baseline CA19-9 in that arm.
Time Frame: First day of treatment to the end of Cycle 2, Week 1
Population: The CA19-9 response rate was calculated for at least the 15 patients in each arm of the study at the end of the first two cycles of therapy (8 weeks) in the mITT population who had elevated CA19-9 levels at baseline.
Measure: Number; unit: Percentage of participants
Arm/Group | Cetuximab + Bevacizumab + Gemcitabine | Cetuximab + Bevacizumab
Number analyzed (Participants) | 18 | 19
Percentage of participants | 8 | 9

5. Secondary Outcome: Time to Progression (TTP)
Description: Time to progression was defined as the time from randomization until the date of objectively confirmed tumor progression was first reported. The censoring rule was consistent with PFS except death. Patients who died from any cause were censored at the time of death or at last tumor assessment date if the death date was missing. For patients lost to follow-up, they were censored at the last tumor assessment date.
Time Frame: Time from randomization until the date of objective tumor progression was first reported (range: 11 -38 months)
Population: The TTP was based on the mITT population. For patients lost to follow-up, they were censored at the next scheduled visit.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cetuximab + Bevacizumab + Gemcitabine | Cetuximab + Bevacizumab
Number analyzed (Participants) | 29 | 29
months | 4.11 [2.17 to 5.95] | 2.07 [1.84 to 4.01]

6. Secondary Outcome: Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: Reported AEs per patient were coded according to the corresponding preferred term and system organ class in the Medical Dictionary for regulatory Activities dictionary. The National Cancer Institute-Common Terminology Criteria for Adverse Events (NCI-CTCAE), Version 3.0 was used to grade all AEs. The collection of AEs began at the time the patient received the first cetuximab dose and continued during the study until 30 days after the last dose of cetuximab. All patients who were enrolled and treated with cetuximab were assessed for safety (mITT population, as treated).
Time Frame: An AE was included in the safety analysis if its onset date occurred anytime during cetuximab treatment or up to 30 days after the last dose of cetuximab.
Population: All patients who received any quantity of study therapy were included in the safety evaluation (safety population, as treated).
Measure: Number; unit: Participants
Arm/Group | Cetuximab + Bevacizumab + Gemcitabine | Cetuximab + Bevacizumab
Number analyzed (Participants) | 29 | 29
Participants | 29 | 29

7. Secondary Outcome: Change From Baseline in Quality of Life (QoL) Assessment Using the Linear Analog Scale Assessment (LASA), Overall QoL at Cycle 2 Week 4
Description: Accrual on the trial was stopped earlier than planned due to insufficient efficacy on both arms. The primary analysis of pancreatic cancer symptoms was conducted using the LASA QoL questionnaire and was considered exploratory. The Overall QoL question change from baseline to Cycle 2 Week 4 is reported. The best overall score is 10 and the worst is 0. A negative score indicates worsening from baseline.
Time Frame: Screening, and then every 8 weeks while receiving study drug to 30-day follow-up
Population: mITT population
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Cetuximab + Bevacizumab + Gemcitabine | Cetuximab + Bevacizumab
Number analyzed (Participants) | 17 | 12
Scores on a scale | -0.9 (2.9) | -0.9 (2.3)

8. Secondary Outcome: Change From Baseline in QoL Assessment Using LASA, Overall Mental Well Being, at Cycle 2 Week 4
Description: Accrual on the trial was stopped earlier than planned due to insufficient efficacy on both arms. The primary analysis of pancreatic cancer symptoms was conducted using the LASA QoL questionnaire and was considered exploratory. The Overall Mental Well Being question change from baseline to Cycle 2 Week 4 is reported. The best overall score is 10 and the worst is 0. A negative score indicates worsening from baseline.
Time Frame: Screening, and then every 8 weeks while receiving study drug to 30-day follow-up
Population: mITT population
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Cetuximab + Bevacizumab + Gemcitabine | Cetuximab + Bevacizumab
Number analyzed (Participants) | 17 | 11
Scores on a scale | 0.6 (2.0) | -0.8 (1.4)

9. Secondary Outcome: Change From Baseline in QoL Assessment Using LASA, Overall Physical Well Being, at Cycle 2 Week 4
Description: Accrual on the trial was stopped earlier than planned due to insufficient efficacy on both arms. The primary analysis of pancreatic cancer symptoms was conducted using the LASA QoL questionnaire and was considered exploratory. The Overall Physical Well Being question change from baseline to Cycle 2 Week 4 is reported. The best overall score is 10 and the worst is 0. A negative score indicates worsening from baseline.
Time Frame: Screening, and then every 8 weeks while receiving study drug to 30-day follow-up
Population: mITT population
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Cetuximab + Bevacizumab + Gemcitabine | Cetuximab + Bevacizumab
Number analyzed (Participants) | 17 | 12
Scores on a scale | -0.6 (3.1) | -0.6 (1.7)

10. Secondary Outcome: Change From Baseline in QoL Assessment Using LASA, Overall Emotional Well Being, at Cycle 2 Week 4
Description: Accrual on the trial was stopped earlier than planned due to insufficient efficacy on both arms. The primary analysis of pancreatic cancer symptoms was conducted using the LASA QoL questionnaire and was considered exploratory. The Overall Emotional Well Being question change from baseline to Cycle 2 Week 4 is reported. The best overall score is 10 and the worst is 0. A negative score indicates worsening from baseline.
Time Frame: Screening, and then every 8 weeks while receiving study drug to 30-day follow-up
Population: mITT Population
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Cetuximab + Bevacizumab + Gemcitabine | Cetuximab + Bevacizumab
Number analyzed (Participants) | 17 | 11
Scores on a scale | -0.2 (2.8) | -1.1 (2.1)

11. Secondary Outcome: Change From Baseline in QoL Assessment Using LASA, Level of Social Activity, at Cycle 2 Week 4
Description: Accrual on the trial was stopped earlier than planned due to insufficient efficacy on both arms. The primary analysis of pancreatic cancer symptoms was conducted using the LASA QoL questionnaire and was considered exploratory. The Level of Social Activity question change from baseline to Cycle 2 Week 4 is reported. The best overall score is 10 and the worst is 0. A negative score indicates worsening from baseline.
Time Frame: Screening, and then every 8 weeks while receiving study drug to 30-day follow-up
Population: mITT population
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Cetuximab + Bevacizumab + Gemcitabine | Cetuximab + Bevacizumab
Number analyzed (Participants) | 17 | 12
Scores on a scale | -1.1 (2.9) | 0.6 (2.3)

12. Secondary Outcome: Change From Baseline in QoL Assessment Using LASA, Overall Spiritual Well Being, at Cycle 2 Week 4
Description: Accrual on the trial was stopped earlier than planned due to insufficient efficacy on both arms. The primary analysis of pancreatic symptoms was conducted using the LASA QoL questionnaire and was considered exploratory. The Overall Spiritual Well Being question change from baseline to Cycle 2 Week 4 is reported. The best overall score is 10 and the worst is 0. A negative score indicates worsening from baseline.
Time Frame: Screening, and then every 8 weeks while receiving study drug to 30-day follow-up while receiving study drug
Population: mITT population
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Cetuximab + Bevacizumab + Gemcitabine | Cetuximab + Bevacizumab
Number analyzed (Participants) | 17 | 11
Scores on a scale | -0.4 (1.8) | -0.3 (1.1)

13. Secondary Outcome: Change From Baseline in QoL Assessment Using LASA, Frequency of Pain, at Cycle 2 Week 4
Description: Accrual on the trial was stopped earlier than planned due to insufficient efficacy on both arms. The primary analysis of pancreatic cancer symptoms was conducted using the LASA QoL questionnaire and was considered exploratory. The Frequency of Pain question change from baseline to Cycle 2 Week 4 is reported. The best overall score is 10 and the worst is 0. A negative score indicates improvement from baseline.
Time Frame: Screening, and then every 8 weeks while receiving study drug to 30-day follow-up
Population: mITT population
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Cetuximab + Bevacizumab + Gemcitabine | Cetuximab + Bevacizumab
Number analyzed (Participants) | 17 | 12
Scores on a scale | -1.5 (2.9) | -2.3 (2.6)

14. Secondary Outcome: Change From Baseline in QoL Assessment Using LASA, Severity of Pain, Average, at Cycle 2 Week 4
Description: Accrual on the trial was stopped earlier than planned due to insufficient efficacy on both arms. The primary analysis of pancreatic cancer symptoms was conducted using the LASA QoL questionnaire and was considered exploratory. The Severity of Pain question change from baseline to Cycle 2 Week 4 is reported. The best overall score is 10 and the worst is 0. A positive score indicates improvement from baseline.
Time Frame: Screening, and then every 8 weeks while receiving study drug to 30-day follow-up while receiving study drug
Population: mITT population
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Cetuximab + Bevacizumab + Gemcitabine | Cetuximab + Bevacizumab
Number analyzed (Participants) | 17 | 12
Scores on a scale | -0.5 (2.8) | -0.9 (2.4)

15. Secondary Outcome: Change From Baseline in QoL Assessment Using LASA, Level of Fatigue, Average, at Cycle 2 Week 4
Description: Accrual on the trial was stopped earlier than planned due to insufficient efficacy on both arms. The primary analysis of pancreatic cancer symptoms was conducted using the LASA QoL questionnaire and was considered exploratory. The Level of Fatigue question change from baseline to Cycle 2 Week 4 is reported. The best overall score is 10 and the worst is 0. A positive score indicates improvement from baseline.
Time Frame: Screening, and then every 8 weeks while receiving study drug to 30-day follow-up
Population: mITT Population
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Cetuximab + Bevacizumab + Gemcitabine | Cetuximab + Bevacizumab
Number analyzed (Participants) | 17 | 12
Scores on a scale | 1.5 (2.3) | 0.3 (2.6)

16. Secondary Outcome: Change From Baseline in QoL Assessment Using LASA, Level of Support, Friends and Family, at Cycle 2 Week 4
Description: Accrual on the trial was stopped earlier than planned due to insufficient efficacy on both arms. The primary analysis of pancreatic cancer symptoms was conducted using the LASA QoL questionnaire and was considered exploratory. The Level of Support, Friends and Family question change from baseline to Cycle 2 Week 4 is reported. The best overall score is 10 and the worst is 0. A negative score indicates worsening from baseline.
Time Frame: Screening, and then every 8 weeks while receiving study drug to 30-day follow-up
Population: mITT Population
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Cetuximab + Bevacizumab + Gemcitabine | Cetuximab + Bevacizumab
Number analyzed (Participants) | 17 | 12
Scores on a scale | 0.1 (1.3) | -0.8 (1.5)

17. Secondary Outcome: Change From Baseline in QoL Assessment Using LASA, Financial Concerns, at Cycle 2 Week 4
Description: Accrual on the trial was stopped earlier than planned due to insufficient efficacy on both arms. The primary analysis of pancreatic cancer symptoms was conducted using the LASA QoL questionnaire and was considered exploratory. The Financial Concerns Question question change from baseline to Cycle 2 Week 4 is reported. The best overall score is 10 and the worst is 0. A negative score indicates worsening from baseline.
Time Frame: Screening, and then every 8 weeks while receiving study drug to 30-day follow-up
Population: mITT population
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Cetuximab + Bevacizumab + Gemcitabine | Cetuximab + Bevacizumab
Number analyzed (Participants) | 17 | 12
Scores on a scale | -0.1 (2.4) | 0.9 (3.7)

18. Secondary Outcome: Change From Baseline in QoL Assessment Using LASA, Legal Concerns, at Cycle 2 Week 4
Description: Accrual on the trial was stopped earlier than planned due to insufficient efficacy on both arms. The primary analysis of pancreatic cancer symptoms was conducted using the LASA QoL questionnaire and was considered exploratory. The Legal Concerns question change from baseline to Cycle 2 Week 4 is reported. The best overall score is 10 and the worst is 0. A negative score indicates worsening from baseline.
Time Frame: Screening, and then every 8 weeks while receiving study drug to 30-day follow-up
Population: mITT population
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Cetuximab + Bevacizumab + Gemcitabine | Cetuximab + Bevacizumab
Number analyzed (Participants) | 17 | 12
Scores on a scale | 0.4 (1.7) | 2.3 (3.2)

19. Secondary Outcome: Change From Baseline in Assessment of Pain Using the Brief Pain Inventory (BPI) Short Form, Worst Pain, at Cycle 2 Week 4
Description: Accrual on the trial was stopped earlier than planned due to insufficient efficacy on both arms. Analysis of pain using the BPI was considered exploratory. The Worst Pain (change from baseline) to Cycle 2 Week 4 is reported. The worst pain is 10 and no pain is 0. A negative score indicates improvement from baseline.
Time Frame: Screening, and then every 8 weeks while receiving study drug to 30-day follow-up
Population: mITT population
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Cetuximab + Bevacizumab + Gemcitabine | Cetuximab + Bevacizumab
Number analyzed (Participants) | 17 | 12
Scores on a scale | -1.2 (2.8) | 0.5 (2.5)

20. Secondary Outcome: Change From Baseline in Assessment of Pain Using BPI Short Form, Least Pain, at Cycle 2 Week 4
Description: Accrual on the trial was stopped earlier than planned due to insufficient efficacy on both arms. Analysis of pain using the BPI was considered exploratory. The Least Pain (change from baseline) to Cycle 2 Week 4 is reported. The worst pain is 10 and no pain is 0. A negative score indicates improvement from baseline.
Time Frame: Screening, and then every 8 weeks while receiving study drug to 30-day follow-up
Population: mITT population
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Cetuximab + Bevacizumab + Gemcitabine | Cetuximab + Bevacizumab
Number analyzed (Participants) | 17 | 12
Scores on a scale | -0.4 (2.0) | 0.9 (2.4)

21. Secondary Outcome: Change From Baseline in Assessment of Pain Using BPI Short Form, Average Pain, at Cycle 2 Week 4
Description: Accrual on the trial was stopped earlier than planned due to insufficient efficacy on both arms. Analysis of pain using the BPI was considered exploratory. The Average Pain (change from baseline) to Cycle 2 Week 4 is reported. The worst pain was 10 and no pain is 0. A negative score indicates improvement from baseline.
Time Frame: Screening, and then every 8 weeks while receiving study drug to 30-day follow-up
Population: mITT population
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Cetuximab + Bevacizumab + Gemcitabine | Cetuximab + Bevacizumab
Number analyzed (Participants) | 17 | 12
Scores on a scale | -0.6 (1.8) | -0.2 (2.1)

22. Secondary Outcome: Change From Baseline in Assessment of Pain Using BPI Short Form, Pain Right Now, at Cycle 2 Week 4
Description: Accrual on the trial was stopped earlier than planned due to insufficient efficacy on both arms. Analysis of pain using the BPI was considered exploratory. The Pain Right Now question (change from baseline) to Cycle 2 Week 4 is reported. The worst pain is 10 and no pain is 0. A negative score indicates improvement from baseline.
Time Frame: Screening, and then every 8 weeks while receiving study drug to 30-day follow-up
Population: mITT population
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Cetuximab + Bevacizumab + Gemcitabine | Cetuximab + Bevacizumab
Number analyzed (Participants) | 17 | 12
Scores on a scale | -0.9 (2.6) | 0.9 (2.0)

23. Secondary Outcome: Change From Baseline in Assessment of Pain Using BPI Short Form, Interference, at Cycle 2 Week 4
Description: Accrual on the trial was stopped earlier than planned due to insufficient efficacy on both arms. Analysis of pain using the BPI was considered exploratory. The Interference question (change from baseline) to Cycle 2 Week 4 is reported. Complete interference is scored as 10 and no interference is scored as 0. A negative score indicates improvement from baseline.
Time Frame: Screening, and then every 8 weeks while receiving study drug to 30-day follow-up
Population: mITT population
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Cetuximab + Bevacizumab + Gemcitabine | Cetuximab + Bevacizumab
Number analyzed (Participants) | 16 | 12
Scores on a scale | -0.2 (2.3) | 0.8 (2.9)

ADVERSE EVENTS:
Time Frame: Adverse events were collected beginning at the time the patient received the initial cetuximab infusion and continued throughout the study until 30 days after the last dose.
Arm/Group | Cetuximab + Bevacizumab + Gemcitabine | Cetuximab + Bevacizumab
Serious Adverse Events (participants affected / at risk) | 21/29 | 16/29
Other Adverse Events (participants affected / at risk) | 29/29 | 29/29
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cetuximab + Bevacizumab + Gemcitabine (N=29) | Cetuximab + Bevacizumab (N=29)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Atrial Fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Cardio-Respiratory Arrest (Cardiac disorders) | 1 (1) | 0 (0)
Abdominal Pain (Gastrointestinal disorders) | 4 (5) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (2) | 3 (3)
Vomiting (Gastrointestinal disorders) | 1 (1) | 4 (4)
Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 1 (2) | 2 (3)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 2 (2)
Upper abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastric outlet obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Disease progression (General disorders) | 5 (5) | 9 (9)
Fatigue (General disorders) | 2 (2) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 1 (1)
Asthenia (General disorders) | 1 (1) | 0 (0)
Death (General disorders) | 1 (1) | 0 (0)
No adverse drug effect (General disorders) | 0 (0) | 1 (1)
Hepatic failure (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hyperbilirubinemia (Hepatobiliary disorders) | 0 (0) | 1 (1)
Portal vein thrombosis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 2 (2) | 1 (1)
Cellulitis (Infections and infestations) | 2 (3) | 0 (0)
Enterococcal sepsis (Infections and infestations) | 1 (1) | 0 (0)
Otitis exterma (Infections and infestations) | 1 (1) | 0 (0)
Pyelonephritis (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 0 (0)
Septic shock (Infections and infestations) | 1 (1) | 0 (0)
Feeding tube complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Overdose (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Stent occlusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Increased alanine aminotransferase (Investigations) | 0 (0) | 1 (1)
Increased aspartate aminotransferase (Investigations) | 0 (0) | 1 (1)
Failure to thrive (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 1 (2) | 1 (1)
Cerebral hemorrhage (Nervous system disorders) | 1 (2) | 0 (0)
Sedation (Nervous system disorders) | 0 (0) | 1 (1)
Acute renal failure (Renal and urinary disorders) | 0 (0) | 2 (2)
Renal failure (Renal and urinary disorders) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 2 (2)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Acneiform dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 2 (2) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 2 (2)
Arterial occlusive disease (Vascular disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cetuximab + Bevacizumab + Gemcitabine (N=29) | Cetuximab + Bevacizumab (N=29)
Anemia (Blood and lymphatic system disorders) | 9 (23) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 9 (21) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 9 (22) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 3 (6) | 0 (0)
Tachycardia (Cardiac disorders) | 1 (1) | 2 (2)
Cardiomegaly (Cardiac disorders) | 2 (2) | 0 (0)
Nausea (Gastrointestinal disorders) | 14 (19) | 14 (20)
Vomiting (Gastrointestinal disorders) | 11 (17) | 9 (12)
Constipation (Cardiac disorders) | 11 (12) | 7 (7)
Stomatitis (Gastrointestinal disorders) | 9 (13) | 7 (8)
Diarrhea (Gastrointestinal disorders) | 9 (10) | 4 (4)
Abdominal pain (Gastrointestinal disorders) | 4 (6) | 2 (2)
Abdominal distention (Gastrointestinal disorders) | 2 (2) | 3 (3)
Upper abdominal pain (Gastrointestinal disorders) | 3 (3) | 2 (2)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 4 (4)
Oral pain (Gastrointestinal disorders) | 2 (2) | 2 (2)
Flatulence (Gastrointestinal disorders) | 2 (2) | 0 (0)
Hemorrhoids (Gastrointestinal disorders) | 2 (2) | 0 (0)
Fatigue (General disorders) | 20 (32) | 10 (13)
Pyrexia (General disorders) | 8 (9) | 3 (3)
Peripheral edema (General disorders) | 7 (11) | 3 (5)
Chills (General disorders) | 4 (5) | 3 (3)
Infusion related reaction (General disorders) | 3 (4) | 2 (2)
Pain (General disorders) | 2 (2) | 3 (3)
Asthenia (General disorders) | 2 (2) | 0 (0)
Malaise (General disorders) | 2 (2) | 0 (0)
Jaundice (Hepatobiliary disorders) | 3 (3) | 2 (2)
Bile duct obstruction (Hepatobiliary disorders) | 2 (2) | 0 (0)
Hyperbilirubinemia (Hepatobiliary disorders) | 2 (2) | 0 (0)
Cholestatic jaundice (Hepatobiliary disorders) | 2 (2) | 0 (0)
Urinary tract infection (Infections and infestations) | 4 (4) | 2 (2)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 2 (2)
Anorexia (Metabolism and nutrition disorders) | 13 (19) | 9 (12)
Dehydration (Metabolism and nutrition disorders) | 4 (4) | 6 (8)
Hypomagnesemia (Metabolism and nutrition disorders) | 7 (12) | 3 (3)
Hypokalemia (Metabolism and nutrition disorders) | 5 (11) | 3 (3)
Hyperglycemia (Metabolism and nutrition disorders) | 2 (3) | 2 (2)
Hyperkalemia (Metabolism and nutrition disorders) | 3 (3) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Hypermagnesemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Hypocalcemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Extremity pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 3 (4) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Headache (Nervous system disorders) | 6 (14) | 5 (5)
Dizziness (Nervous system disorders) | 5 (5) | 1 (1)
Dysgeusia (Nervous system disorders) | 3 (3) | 2 (2)
Depression (Psychiatric disorders) | 5 (6) | 4 (4)
Anxiety (Psychiatric disorders) | 3 (3) | 4 (4)
Insomnia (Psychiatric disorders) | 4 (4) | 2 (2)
Confusional state (Psychiatric disorders) | 1 (2) | 2 (2)
Mental Disorder (Psychiatric disorders) | 0 (0) | 2 (2)
Proteinuria (Renal and urinary disorders) | 6 (7) | 2 (2)
Acute renal failure (Renal and urinary disorders) | 2 (2) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 8 (10) | 4 (4)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 3 (3)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
Exertional dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Acneiform dermatitis (Respiratory, thoracic and mediastinal disorders) | 22 (48) | 21 (27)
Pruritus (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 2 (2)
Skin disorder (Skin and subcutaneous tissue disorders) | 1 (2) | 5 (5)
Dry skin (Skin and subcutaneous tissue disorders) | 4 (4) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 2 (2) | 3 (4)
Alopecia (Skin and subcutaneous tissue disorders) | 4 (4) | 0 (0)
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 4 (5) | 1 (1)
Hypertension (Vascular disorders) | 2 (2) | 2 (3)
Hypotension (Vascular disorders) | 2 (2) | 1 (1)

LIMITATIONS AND CAVEATS:
Accrual on the trial was stopped earlier than planned due to insufficient efficacy in both arms.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Investigators agreed to delay independently publishing or disclosing data, findings or conclusions from the study except as part of a multi-center publication. Upon study publication or if draft publication is not produced within approximately 6 months of the final report of the study results, investigators may independently publish, subject to confidential information review/redaction by sponsor. Sponsor may request publication delay up to 90 days to seek patent protection.